CLINICAL TRIAL: NCT01061203
Title: Grazax Asthma Prevention
Acronym: GAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GT-21
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Allergic Rhinitis
Keywords: Rhinitis; allergic; Seasonal; grass; Asthma
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis; Asthma | interventions — Grazax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grazax (Active Comparator): Grazax tablet 75.000 SQ-T. One tablet per day for administration under the tongue.
  Interventions: Drug: Grazax
- Tablet with no active grass (Placebo Comparator): Tablet with no active grass component. One tablet per day administered under the tongue.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Grazax — Treatment with 75.000 SQ-T once daily
  Arms: Grazax
Drug: Placebo — Tablet with no active grass component.
  Arms: Tablet with no active grass

SUMMARY:
Investigation of the effect of Grazax (grass tablet) on asthma prevention in children with grass pollen allergy

DETAILED DESCRIPTION:
Investigation of the effect of Grazax (ALK produced grass tablet) on asthma prevention in children with grass pollen allergy.

Children in the age of 6-12 years will be randomised to either placebo or Grazax treatment. Grazax has been approved for treatment of grass pollen allergy in adults and children, diagnosed with a positive skin prick test and/or specific immunoglobulin (IgE) test to grass pollen and with clinically relevant symptoms. This study will explore prevention of asthma in children with grass pollen induced allergy.

ELIGIBILITY:
Inclusion Criteria:

* A history of grass pollen allergy
* Positive Skin prick test to grass
* Positive specific IgE to grass

Exclusion Criteria:

* Asthma

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 812 (Actual)
Dates: Start 2010-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of allergy and asthma symptoms | 5 years

SECONDARY OUTCOMES:
Quality of life and adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Erkka Valovirta, MD, Principal Investigator — Terveystalo Turku, Finland
Locations (1):
- Terveystalo Turku, Turku, Finland